CLINICAL TRIAL: NCT00339807
Title: Natural History of HTVL-I: A Cross-Sectional Study of a Cohort of Blood Donors in Jamaica
Brief Title: Natural History of HTLV-I Infection: Prospective Follow-up of a Cohort of Blood Donors in Jamaica
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902112; 02-C-N112; NCT00544661 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-11

CONDITIONS: HTLV-I
Keywords: Retrovirus; Caribbean; Transmission; Genetic; Viral Markers; HTLV-1

SUMMARY:
Human T-lymphotrophic virus type I (HTLV-I) is endemic in southern Japan and the Caribbean, but disease manifestations differ across geographic regions. Though age, gender, and route of infection may determine the natural history of this infection, the observed geographic differences also may, in part, reflect the distinct genetic background of the host as evidenced by the distribution of human leukocyte antigens (HLA) and the presence of other environmental factors.

Studies already completed or ongoing have shown notable differences in incidence and prevalence of HTLV-I associated diseases and underscore the need for comparative studies and analyses in these areas. This prospective new study of blood donors in Jamaica provides us with an opportunity to address many hypotheses regarding HTLV-I transmission and pathogenesis in the Caribbean in comparison with an ongoing cohort study of HTLV-I carriers in Japan.

This study will

* identify host factors associated with HTLV-I carrier status and HTLV-I pathogenesis.
* directly calculate the incidence of HTLV-I associated diseases in this population.
* examine the role of HTLV-I in the pathogenesis of other common infectious agents.

Approximately 5,000+ blood donors who came to the National Blood Transfusion each year will be screened for HTLV-I serology. Of those who agreed to participate, all HTLV-I carriers and age-, and sex-matched HTLV-I-negatives will be invited to the University of the West Indies clinic for a full study enrollment. Study participants will be given a standardized questionnaire, a full physical examination, and a phlebotomy (25-30 mL), and will be followed every other year for interim health status and additional phlebotomy. All subjects will receive an ophthalmologic examination for detection of uveitis and other ocular diseases. Some subjects will be further referred to a neurologist, hematologist or dermatologist, according to their signs and symptoms. Approximately 1200 HTLV-I carriers and 600 HTLV-I negatives will be recruited for a longitudinal follow-up over the next 5-year period. Two types of analyses will be conducted: comparison of HTLV-I-positive and HTLV-I-negative subjects, and comparison among HTLV carriers between those with a high level of viral load and those with a low level.

DETAILED DESCRIPTION:
Southern Japan and the Caribbean are both endemic for human T-lymphotropic virus type I (HTLV-I) infection. In these areas, however, epidemiology of HTLV-I appears to differ. Various observations from population-based studies indicate that differences in host immune response to virus infection is likely to result in different frequencies of disease manifestations across geographic regions. While gender, age and route of infection may partly determine host immune response, the observed geographic differences may also reflect, in part, host genetic background as evidenced by the distribution of human leukocyte antigens (HLA) and presence of other environmental factors.

The reported differences underscore the need for comparative studies in these endemic areas. In addition, analyses of larger, pooled data of HTLV-I carriers from different geographic areas are needed to ensure statistical power in studies of gene-environment interactions with extended use of molecular markers. However, existing population-based studies from Japan and the Caribbean are unfortunately no comparable with respect to the study subject's age and gender distributions. In order to address this issue, we proposed a study of blood donors in Jamaica, which enrolls a large number of both HTLV-I positive and HTLV-I negative, consisting of subjects that are more comparable to existing Japanese study with respect to age and sex. The proposed study will provide a basis for a comparative study of HTLV-I carriers in Japan and Jamaica and a comprehensive analysis of host genetic background of HTLV-I associated illnesses in the Black population.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy blood donors in Kingston, Jamaica.

All HTLV-I positive donors and age-, sex-matched HTLV-1 negative donors (controls) will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2002-01-17; Study Completion 2011-08-11

CONTACTS AND LOCATIONS:
Locations (1):
- University of the West Indies, Kingston, Jamaica

REFERENCES:
- [Background] Poiesz BJ, Ruscetti FW, Gazdar AF, Bunn PA, Minna JD, Gallo RC. Detection and isolation of type C retrovirus particles from fresh and cultured lymphocytes of a patient with cutaneous T-cell lymphoma. Proc Natl Acad Sci U S A. 1980 Dec;77(12):7415-9. doi: 10.1073/pnas.77.12.7415. PMID 6261256
- [Background] Hinuma Y, Nagata K, Hanaoka M, Nakai M, Matsumoto T, Kinoshita KI, Shirakawa S, Miyoshi I. Adult T-cell leukemia: antigen in an ATL cell line and detection of antibodies to the antigen in human sera. Proc Natl Acad Sci U S A. 1981 Oct;78(10):6476-80. doi: 10.1073/pnas.78.10.6476. PMID 7031654
- [Background] Madeleine MM, Wiktor SZ, Goedert JJ, Manns A, Levine PH, Biggar RJ, Blattner WA. HTLV-I and HTLV-II world-wide distribution: reanalysis of 4,832 immunoblot results. Int J Cancer. 1993 May 8;54(2):255-60. doi: 10.1002/ijc.2910540216. PMID 8486428